CLINICAL TRIAL: NCT02981927
Title: Bed Rest, Inactivity and Early Responses
Acronym: BIER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 157758/02
Record Dates: First submitted 2016-11-30; First posted 2016-12-05 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Metabolic Responses to Inactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): 24 h habitual physical activity fed in energy balance
- Bed rest matched diet (Experimental): 24 hour period of whole body bed-rest with a matched diet
  Interventions: Other: Physical inactivity
- Bed rest balanced diet (Experimental): 24 hour period of whole body bed-rest fed in energy balance
  Interventions: Other: Physical inactivity

INTERVENTIONS:
Other: Physical inactivity
  Arms: Bed rest balanced diet; Bed rest matched diet

SUMMARY:
To evaluate the early metabolic responses (whole body and within muscle tissue) to a single day of whole body physical inactivity (i.e. bed-rest), and evaluate the contribution of inactivity per se vs alterations in diet

ELIGIBILITY:
Inclusion Criteria:

* Healthy and aged 18-40 y
* BMI between 18 and 30

Exclusion Criteria:

* On medication
* Family history of metabolic disease
* Diagnosed with any metabolic or cardiovascular conditions
* BMI < 18 or > 30

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12-02 (Actual); Study Completion 2016-12-02 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Sport & Health Sciences, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No